CLINICAL TRIAL: NCT02446145
Title: A Randomized Placebo-controlled Phase 2 Study of Decitabine With or Without Eltrombopag in AML Patients ≥65 Years of Age Not Eligible for Intensive Chemotherapy
Brief Title: A Randomized Placebo-controlled Phase 2 Study of Decitabine With or Without Eltrombopag in AML Patients
Acronym: DELTA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to COVID-19 pandemia, recruitment was insufficient to reach required sample size in an acceptable time line. Furthermore, new drugs have recently been licensed resulting in alternative treatment regimens with a better prognosis.
Sponsor: Technische Universität Dresden (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TUD-DELTA1-063; 2014-003150-13 (EudraCT Number)
Record Dates: First submitted 2015-02-11; First posted 2015-05-18 (Estimated); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental intervention arm (Experimental): Eltrombopag daily from day 12 to 25: 200 mg/day p.o. (100 mg for east asian patients) dose modification 100 mg up to 300 mg/d p.o. (50 - 150 mg for east asian patients)
  * concomitant medication: either Decitabine days 1-5 of each cycle: 20 mg/sqm i.v. over 30 minutes or Azacitidine (AZA) days 1-7 of each cycle: 75 mg/sqm s.c.
  * one cycle lasts 28 days
  Interventions: Drug: Eltrombopag
- Control intervention arm (Placebo Comparator): Placebo daily from day 1: 200 mg/day p.o. (100 mg for east asian patients) dose modification 100 mg up to 300 mg/d p.o. (50 - 150 mg for east asian patients)
  * concomitant medication: either Decitabine days 1-5 of each cycle: 20 mg/sqm i.v. over 30 minutes or Azacitidine (AZA) days 1-7 of each cycle: 75 mg/sqm s.c.
  * one cycle lasts 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eltrombopag — Patients will receive EPAG in addition to their background standard treatment with Decitabine/Azacitidine
  - concomitant medication: either Decitabine days 1-5 of each cycle: 20 mg/sqm i.v. over 30 minutes or Azacitidine (AZA) days 1-7 of each cycle: 75 mg/sqm s.c.
  Other Names: Revolade
  Arms: Experimental intervention arm
Drug: Placebo — Patients will receive Placebo in addition to their background standard treatment with Decitabine/Azacitidine
  - concomitant medication: either Decitabine days 1-5 of each cycle: 20 mg/sqm i.v. over 30 minutes or Azacitidine (AZA) days 1-7 of each cycle: 75 mg/sqm s.c.
  Arms: Control intervention arm

SUMMARY:
Acute myeloid leukemia (AML) is a disease with a poor prognosis including a 5-year overall survival (OS) of app. 20% for the entire population. In particular, the outcome of elderly patients with AML is dismal and the majority of patients die within the first year after diagnosis. This is also because treatment options for elderly patients with AML significantly differ from patients of younger age. In fact, comorbid conditions are common among the elderly such as heart disease, renal insufficiency and vascular disease thus influencing the ability to withstand intensive therapy. Elderly patients are also more likely than younger patients to develop severe, life threatening infections during the course of treatment. In addition to infectious complications, hemorrhages due to severe thrombocytopenia are responsible for morbidity and mortality in a considerable amount of patients. Compared with younger AML patients, elderly individuals with AML display a higher incidence of poor-prognosis karyotypes, of a preceding myelodysplastic syndrome (MDS), and greater expression of proteins involved in intrinsic resistance to chemotherapeutic agents. As a result conventional anthracycline based chemotherapy is only infrequently used in patients above the age of 65 years. Based on a recent randomized trial (Kantarjian et al. 2012) low-intensity epigenetic therapy with decitabine (DAC) has become the first-line standard of care in most European countries including Germany. Nevertheless, even with this treatment the 1-year OS is approximately 30 % only. Furthermore, severe thrombocytopenia is a main side effect of this therapy and can prevent adequate continuation of treatment being crucially for treatment success. Supportive care with platelet transfusions is effective primarily only over short periods and often requires hospitalization and therefore lowers the quality of life of these patients in their palliative situation. Therefore, patients could benefit from an approach aiming at an increase of platelet counts through combined use of Azacitidine (AZA) or DAC with an oral thrombopoietin receptor agonist like eltrombopag (EPAG). This could allow for a better adherence to DAC/AZA therapy by preventing dose delays due to prolonged thrombocytopenia. Additionally, the potential antileukemic effect of EPAG could also be beneficial for these AML patients.

DETAILED DESCRIPTION:
The DELTA-trial is designed as a two-arm, double-blind, multicenter randomized-controlled phase- II study of EPAG or placebo in combination with standard-dose DAC/AZA treatment as concomitant medication in subjects at least 65 years of age with AML not eligible for intensive chemotherapy and planned therapy with Decitabine (DAC)/Azacitidine(AZA). Patients will be randomized 1:1 into the experimental study arm and the control study arm. EPAG 200 mg (100 mg for East Asian patients) once daily has been selected as the starting dose for this study because this regimen has been investigated to be safe and potentially effective in increasing platelet counts in patients with AML. Concomitant medication with DAC/AZA will be according to the european label and the summary of product characteristics. There will be a dose adjustment of EPAG depending on the platelet counts obtained on day 1 of a planned DAC/AZA cycle. EPAG or placebo will be taken for 14 days in each treatment cycle starting on day 12 with a minimum treatment gab of 2 days before and after each DAC/AZA course.

Concomitant medication will be either Decitabine (DAC) 20 mg/m2 body surface i.v. over 30 minutes on days 1-5 of each cycle or Azacitidine (AZA) 75 mg/m2 body surface sc. on days 1-7. One cycle lasts 28 days.

Patients will receive medication as long as they benefit from treatment and in the absence of relevant adverse events indicating a treatment discontinuation; but for a maximum of 12 cycles. During Follow Up (up to 4 years) patient survival and first treatment change will be observed.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AML (including therapy-related or with antecedent MDS) other than acute promyelocytic leukemia (APL) according to WHO criteria, i.e. bone marrow aspirate / biopsy or peripheral blood must contain ≥20% blasts in AML defined by cytogenetic aberrations according to WHO the proportion of blasts may be <20%
* Age ≥ 65 years
* Eastern Cooperative Oncology Group performance status (ECOG) 0-3
* patients not eligible for intensive induction therapy (according to investigator's decision)
* planned therapy with DAC/AZA
* platelet count <75 Gpt/L taken within 4 weeks prior to randomization
* adequate liver function as assessed by the following laboratory requirements during screening (within 4 weeks prior to study inclusion):

  * Total bilirubin ≤ 3 times the upper limit of normal (except for Gilbert's Syndrome)
  * Alanine transaminase (ALAT) and Aspartate transaminase (ASAT) ≤ 3 times upper limit of normal
* signed Informed Consent

Exclusion Criteria:

* acute promyelocytic leukemia (APL)
* history of higher-risk MDS or AML treatment with thrombopoietin receptor (TPO-R) agonists, hypomethylating agents or intensive chemotherapy
* substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* treatment with an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding to first dose of study mediation
* uncontrolled active infection
* New York Heart Association (NYHA) stage ≥ 2 due to heart insufficiency
* positive Human Immunodeficiency Virus (HIV) or Hepatitis B / C serology
* patients unable to swallow medication
* known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to EPAG or DAC or excipients that contraindicates their participation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 132 (Actual)
Dates: Start 2015-05; Primary Completion 2020-12-26 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
treatment change-free survival | up to 4 years
  time from randomization until day one of the new disease modifying treatment or death as the primary endpoint of this study

SECONDARY OUTCOMES:
overall survival | up to 4 years
  Overall survival is defined as months from day 1 of cycle 1 until death and is calculated as (date of death - date of day 1 of cycle 1 + 1) / 30.43
relapse free survival | up to 4 years
  Relapse free survival is defined for patients who achieved CR, CRi, CRc, or CRm.
overall response rate | up to 4 years
  Overall response is defined as achievement of stable disease (SD), partial remission (PR), or complete remission (CR, including CRi, CRc, CRm) at any time during treatment period.
number of bone marrow blasts after 5, 9, and 12 months | screening, month 5, 9 and 12
  Bone marrow blasts are determined locally and by central review. The blast count from the central review is preferred in the analysis. In case of missing blast count from central review the locally determined blast count will be used for analysis.
quality of life questionnaire (QLQ-C30) | screening, month 1, 3, 6, 9, 12
  Quality of life is assessed by the EORTC QLQ-C30 and the SF36 questionnaires. Quality of life will be assessed only in patients with complete baseline assessment. QOL will only be assessed in analysis sets for which information is available for more than 75% of individuals.
Short Form questionnaire 36 (SF-36) | screening, month 1, 3, 6, 9, 12
  Quality of life is assessed by the EORTC QLQ-C30 and the SF36 questionnaires. Quality of life will be assessed only in patients with complete baseline assessment. QOL will only be assessed in analysis sets for which information is available for more than 75% of individuals.
median platelet counts | month 1 - 12
  Platelet counts are analysed as recorded in the study database.
number of platelet transfusions | month 1 - 4
  Number of platelet transfusions during cycle 1-4 is defined as the cumulative sum of platelet transfusions documented in cycles 1 to 4.
incidence of serious adverse events (SAE) | up to 4 years
  incidence of SAE including death, incidence of bleeding events and hospitalization rate and duration

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Platzbecker, Prof., Principal Investigator — Universitätsklinikum Dresden Medizinische Klinik und Poliklinik I
Locations (15):
- Germany (15):
  - Uniklinik RWTH Aachen, Aachen
  - Charite Campus Benjamin Franklin, Berlin
  - Klinikum Chemnitz GmbH, Chemnitz
  - Universitätsklinikum Dresden, Dresden
  - Marienhospital Düsseldorf GmbH, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Halle (Saale), Halle
  - St. Marien-Hospital Hamm, Hamm
  - Klinikum rechts der Isar der TU München, München
  - Klinikum Nürnberg-Nord, Nuremberg
  - Medizinisches Versorgungszentrum für Blut- und Krebserkrankungen, Potsdam
  - Wissenschaftskontor Nord GmbH & Co KG, Rostock
  - Diakonie-Klinikum Schwäbisch Hall gGmbH, Schwäbisch Hall
  - Rems-Murr-Klinikum Winnenden, Winnenden
  - Universitätsklinikum Würzburg, Würzburg

REFERENCES:
- See also: homepage of study group — http://www.sal-aml.org